CLINICAL TRIAL: NCT03273049
Title: Coordinating Center- Mapping Disease Pathways for Biliary Atresia
Brief Title: Mapping Disease Pathways for Biliary Atresia
Acronym: BA
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rakesh Sindhi, Rakesh Sindhi, MD, Professor of Surgery, University of Pittsburgh
Other Study IDs: STUDY19070273; 1R01DK109365-01A1 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA: blood, saliva or liver tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will primarily evaluate the developmental/genetic basis of biliary atresia, the most common cause of liver failure at birth, and which accounts of half of all liver transplants performed worldwide in children.

DETAILED DESCRIPTION:
Characterized by failure to drain bile from the liver due to atretic extrahepatic bile ducts, BA is corrected in less than half of all affected children with surgical reconstruction. The remainder progress to cirrhosis and require liver transplantation. Because bile duct loss can be accompanied by other birth defects such as laterality defects of the gut and cardiovascular systems, the disease has been categorized into the more common 'isolated' variety presumably due to a perinatal viral cholangitis, and the 'syndromic' variety, due to genetic factors. Mechanistic differences implied by this categorization have not been demonstrated conclusively. In contrast, three susceptibility genes identified in predominantly 'isolated" BA cases, and the presence of abnormal cilia which are known to predispose to laterality defects, in both isolated and syndromic forms of BA suggest that in addition to environmental influences, genetic susceptibility is important in both forms of BA. This view is reinforced by our preliminary work which shows that knockdown of a novel BA susceptibility gene causes both biliary dysgenesis and laterality defects in animal models. This finding also suggests that common birth defects affecting the liver and other organs may originate from defects in the same genes. The project will combine candidate gene identification and replication with human DNA samples from 1100 BA subjects and their biological parents or siblings, if available, with validation using corresponding human BA liver tissue and zebrafish knockdown models.

The project outcome will consist of pathways comprising multiple susceptibility genes involved in morphogenesis of the liver and other organs, which explain the complex phenotype of BA. The project will use the experimental and bioinformatics capabilities of the Universities of Pittsburgh and California (at San Diego) to analyze data and study human samples from the participating centers. Four of the world's largest pediatric liver transplant centers, the Children's Hospitals of Pittsburgh (CHP), King's College Hospital (KCH), London, UK, Birmingham Children's Hospital, UK (BCH), and the Hospital Sirio Libanes (HSL), Sao Paulo, Brazil will enroll biliary atresia subjects and their biological parents and/or siblings, if available.

Information developed in this project will be the basis for designing novel management strategies to reduce the societal impact of this rare childhood disease.

ELIGIBILITY:
Inclusion Criteria:

* living individuals who were diagnosed with Biliary Atresia and received or are about to receive a liver transplant from multiple participating centers (Children's Hospital of Pittsburgh, Kings College Hospital, Children's Hospital of Birmingham, and Hospital Sírio-Libanês).

Exclusion Criteria:

* No child participant in the care of the state will be enrolled, nor will patients in the care of temporary or informal guardians be enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have had a liver transplantation due to a diagnosis of biliary atresia.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2030-12-21 (Estimated); Study Completion 2035-07-21 (Estimated)

PRIMARY OUTCOMES:
Genomic pathways of BA | up to two years
  Main project outcome will consist of pathways comprising multiple susceptibility genes involved in morphogenesis of the liver and other organs, which explain the complex phenotype of BA.

SECONDARY OUTCOMES:
Predisposition of BA | upwards of four years to achieve this outcome measure
  determine whether candidate genes and related pathways which predispose to BA, also predispose to laterality defects affecting the liver and other organs.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States